CLINICAL TRIAL: NCT04984395
Title: Improving Diagnosis and Treatment of Metastatic Advanced Prostate Cancer Through Better Imaging With Whole-Body Magnetic Resonance Imaging With Diffusion Weighted Imaging
Brief Title: Improving Diagnosis and Treatment of Metastatic Advanced Prostate Cancer
Acronym: IDT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Royal Marsden NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CCR5459
Record Dates: First submitted 2021-07-21; First posted 2021-07-30 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-05

CONDITIONS: Advanced Prostate Carcinoma

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Bone marrow biopsy.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Post-treatment CT-guided bone marrow biopsy — At post-treatment, 12 +/- 3 weeks after initiating treatment, patients will undergo a CT guided bone marrow biopsy of the same lesion as baseline.

SUMMARY:
The aim of this study is to provide clinical evidence to determine if Whole Body Magnetic Resonance Imaging (WBMRI) with a novel technique called diffusion-weighted imaging (DWI) can improve current treatment for APC patients, allowing for early identification of disease progression or treatment response, hence facilitating clinical decision-making and leading to improvement in patient care. The IDT study includes two retrospective analyses and a single centre prospective observational study for APC patients.

DETAILED DESCRIPTION:
Metastatic Advanced Prostate Cancer occurs when cancer spreads from the prostate to other parts of the body (bones, lymph nodes or other organs), with bones being the commonest site of spread in prostate cancer. These cancer growths are called metastases. APC metastases are diverse (heterogeneous) in their growth pattern, such that not all metastases will respond to the same treatment.

ELIGIBILITY:
Inclusion Criteria:

Retrospective study A Baseline WBMRI scans in metastatic APC patients acquired up to 8 weeks prior to the initiation of a new line of therapy.

Retrospective study B Paired WBMRI scans in metastatic APC patients at baseline within 8 weeks prior to treatment and at 12 ± 3 weeks after systemic treatment

Prospective study C Written informed consent. Age ≥18 years. Advanced prostate cancer patients with indication for systemic anti-cancer therapy to be enrolled in a clinical study.

Participants must have a baseline WBMRI and CT-guided bone marrow biopsy.

Exclusion Criteria:

Prospective Study C Patient is claustrophobic. Contraindications to MRI examination (e.g., cardiac pacemakers, cochlear implants).

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Male with prostate cancer.
Study Population: Patients with metastatic, advanced prostate cancer.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-07-30 (Estimated); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
Retrospective analysis: WBMRI parameters | Month 1-26
  Prognostic association of derived pre-treatment WBMRI parameters, total disease volume (tDV) and apparent diffusion coefficient (ADC) for prediction of overall survival.
Retrospective analysis: Diagnostic performance of MET-RADS-P | Month 1-26
  Accuracy of MET-RADS-P to assess response to systemic treatment.
Single centre prospective observational imaging study | Month 6-38
  Pairwise correlations of percentage of ADC change with:
  1. Tumour regression grading according to the international system of Salzer-Kuntschnik
  2. Changes in biopsy tumour content and tumour/necrosis ratio
  3. Fat fraction percentage with bone marrow adipose tissue/fibrosis reported by histopathology analysis.

SECONDARY OUTCOMES:
Retrospective analysis: WBMRI parameters | Month 1-26
  Prognostic association of baseline tDV and ADC for prediction of radiographic Progression Free Survival (rPFS) using Prostate Cancer Working Group 3 criteria (PCWG3) and Skeletal Related Events (SREs).
Retrospective analysis: Diagnostic performance of MET-RADS-P | Month 1-26
  Inter-observer agreement - determine prognostic association of MET-RADS-P response for prediction of overall survival.
Single centre prospective observational imaging study | Month 6-38
  Fraction of bone biopsies with sufficient tumour yield for genomic sequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Nina Tunariu, Principal Investigator — The Royal Marsden NHS FT
Locations (1):
- The Royal Marsden NHS Foundation Trust, Sutton, Surrey, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
The main study results will be published in a peer-reviewed journal, on behalf of all collaborators. The manuscript will be prepared by a writing group, consisting of members of the Study Management Group.
Supporting Information: CSR
Time Frame: Fully anonymised trial data will be made available.
Access Criteria: Data Sharing / Transfer Agreements to be in place.